CLINICAL TRIAL: NCT04829006
Title: Automatic Assessment of Intelligibility in Individuals With Parkinson's Disease
Brief Title: Intelligibility Assessment for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Long Island University (Other)
Responsible Party: Principal Investigator, Gemma Moya Gale, Assistant Professor, CCC-SLP, Long Island University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21/01-002
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
Keywords: intelligibility; voice disorders; dysarthria
MeSH Terms: conditions — Parkinson Disease; Voice Disorders; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speakers (Other): Participants will be recording sentences using a customized app, which is the focus of the current investigation. There is no arm per se, as the current investigation does not involve an intervention. The current investigation aims at developing and pilot testing an app.
  Interventions: Device: Understand Me For Life

INTERVENTIONS:
Device: Understand Me For Life — The aim of the current investigation is to test the efficacy of an app to measure sentence intelligibility in noise in speakers with Parkinson's disease and in healthy controls.

SUMMARY:
The investigators aim at testing the efficacy of an app to measure sentence intelligibility in noise in speakers with Parkinson's disease and in healthy controls.

DETAILED DESCRIPTION:
Close to 90% of people with Parkinson's disease develop voice problems during the course of the disease. These problems lead to reduced intelligibility, which entails a subsequent reduction in social participation and overall quality of life. The current study will focus on developing and pilot-testing an app to measure the intelligibility of people with PD and of healthy controls. In order to test the app's efficacy, speakers will read a set of 50 sentences that will be embedded in noise for measurement purposes. A group of listeners will also transcribe the spoken sentences to correlate their performance to that of the app. The ultimate purpose of this investigation is to improve self-monitoring and self-sufficiency in people with PD. The study is expected to last 12 months.

ELIGIBILITY:
Speakers with PD:

Inclusion Criteria:

* Have a medical diagnosis of Parkinson's disease
* Have experienced changes in your voice (e.g., your voice has "lost its strength") and your voice is a current concern
* Have not received individual speech therapy for the past 2 years (group therapy is ok)
* Have a stable medication schedule
* Have not received DBS (Deep Brain Stimulation)
* Are a native speaker of American English

Exclusion Criteria:

* If criteria above are not met

Healthy controls:

Inclusion Criteria:

* Be a native speaker of American English
* Have no history of neurological impairment
* Have no history of speech or language problems

Exclusion Criteria:

* If criteria above are not met

Listeners:

Inclusion Criteria:

* Be a native speaker of American English
* Be between 18-55 years old
* Have no history of speech-language-hearing problems
* Pass a free hearing screening
* Have received the Covid19 vaccine

Exclusion Criteria:

* If criteria above are not met

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Transcription scores | 30 minutes
  Percent of words correctly transcribed

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Moya Gale, Ph.D., Principal Investigator — Long Island University
Locations (1):
- Long Island University, Brooklyn, New York, United States